CLINICAL TRIAL: NCT01355224
Title: Communicating Genetic Information for Obesity
Brief Title: Communicating Risk Information for Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Principal Investigator, Catharine Wang, Associate Professor, Boston University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: CW-R21; 1R21HG006073-01 (NIH)
Record Dates: First submitted 2011-05-04; First posted 2011-05-18 (Estimated); Results first posted 2017-03-14 (Actual); Last update posted 2017-03-14 (Actual); Status verified 2017-01

CONDITIONS: Obesity
Keywords: obesity; genetics; risk assessment; health behaviors; randomized controlled trial
MeSH Terms: conditions — Obesity; Health Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- No risk feedback (No Intervention): No obesity risk information given (control)
- Genetic risk feedback (Experimental): Only personal genetic risk information provided
  Interventions: Genetic: Genetic
- Lifestyle risk feedback (Experimental): Only personal lifestyle risk information provided
  Interventions: Behavioral: Lifestyle
- Both genetic or lifestyle risk feedback (Experimental): Personal genetic and lifestyle information provided
  Interventions: Genetic: Genetic; Behavioral: Lifestyle

INTERVENTIONS:
Genetic: Genetic — Relative risk estimates will be presented based on individuals' risk for obesity based on FTO genotype results.
  Other Names: Genetic risk; Genetic risk feedback; FTO gene risk status
  Arms: Both genetic or lifestyle risk feedback; Genetic risk feedback
Behavioral: Lifestyle — Relative risk estimates will be presented based on individuals' risk for obesity due to lifestyle factors.
  Other Names: Lifestyle risk; Lifestyle risk feedback
  Arms: Both genetic or lifestyle risk feedback; Lifestyle risk feedback

SUMMARY:
This study will examine the impact of providing genetic risk information for obesity on people's attitudes and beliefs about obesity, health behaviors and weight outcomes. Specifically, this study will examine the feasibility of using genetic information to motivate efforts to reduce obesity among individuals recruited to the Coriell Personalized Medicine Collaborative (CPMC), see below for description of CPMC.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled feasibility trial to examine the short-term impact of personalized risk feedback for obesity. This study is uniquely situated to provide important data on how individuals interpret various sources of risk information and how they arrive at an overall perception of risk for a condition. Taken altogether, study findings will be used to serve as an overall model for future intervention efforts to effectively communicate obesity risk information with the goal of improving weight management and overall population health.

CPMC-The CPMC is an ongoing evidence-based longitudinal research study designed to determine the utility of using personal genome information in health management and clinical decision-making. They collect saliva samples, perform genetic analysis and provide genetic risk feedback for several disease conditions including coronary artery disease and type 2 diabetes. The present study will build upon the existing genetic testing and web feedback infrastructure at Coriell to conduct behavioral science research to address critical public health questions.

ELIGIBILITY:
Inclusion Criteria:

Must be age 18 or older, active enrollees in the CPMC trial, and able to read and write in English.

Exclusion Criteria:

Individuals that do not meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 798 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catharine Wang, PhD, MSc, Principal Investigator — Boston University
Locations (1):
- Coriell Institute for Medical Research, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data

REFERENCES:
- [Background] Wang C, Gordon ES, Norkunas T, Wawak L, Liu CT, Winter M, Kasper RS, Christman MF, Green RC, Bowen DJ. A randomized trial Examining The Impact Of Communicating Genetic And Lifestyle Risks For Obesity. Obesity (Silver Spring). 2016 Dec;24(12):2481-2490. doi: 10.1002/oby.21661. PMID 27891830
- [Derived] Wang C, Gordon ES, Stack CB, Liu CT, Norkunas T, Wawak L, Christman MF, Green RC, Bowen DJ. A randomized trial of the clinical utility of genetic testing for obesity: design and implementation considerations. Clin Trials. 2014 Feb;11(1):102-13. doi: 10.1177/1740774513508029. Epub 2013 Nov 11. PMID 24216219

RESULTS

PARTICIPANT FLOW:
Groups:
- No Risk Feedback: No risk feedback for obesity was provided.
- Genetic Risk Feedback: FTO variant: Relative risk estimates presented based on individuals' risk for obesity from genotype results.
- Lifestyle Risk Feedback: Lifestyle: Relative risk estimates presented based on individuals' risk for obesity due to personal lifestyle factors (specifically, hours sitting while watching TV).
- Both Genetic and Lifestyle Risk Feedback: FTO variant: Relative risk estimates presented based on individuals' risk for obesity from genotype results.
  Lifestyle: Relative risk estimates presented based on individuals' risk for obesity due to personal lifestyle factors (specifically, hours sitting while watching TV).
Period: Overall Study
Arm/Group | No Risk Feedback | Genetic Risk Feedback | Lifestyle Risk Feedback | Both Genetic and Lifestyle Risk Feedback
Started | 198 | 203 | 196 | 201
Competed Baseline | 191 | 200 | 193 | 193
Completed | 167 | 180 | 177 | 172
Not Completed | 31 | 23 | 19 | 29

BASELINE CHARACTERISTICS:
Population: Based on participants who completed the baseline survey
Groups:
- Total: Total of all reporting groups
Arm/Group | No Risk Feedback | Genetic Risk Feedback | Lifestyle Risk Feedback | Both Genetic and Lifestyle Risk Feedback | Total
Number analyzed (Participants) | 167 | 180 | 177 | 172 | 696
Age, Continuous [Mean (Full Range); unit: years] | 51 [21 to 82] | 51 [20 to 77] | 51 [21 to 81] | 48 [20 to 81] | 50 [20 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 121 | 118 | 122 | 472
  Male | 56 | 59 | 59 | 50 | 224
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 7 | 3 | 15
  Not Hispanic or Latino | 163 | 176 | 170 | 169 | 678
  Unknown or Not Reported | 2 | 1 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 1 | 1 | 6 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 5 | 4 | 5 | 16
  White | 155 | 166 | 161 | 154 | 636
  More than one race | 2 | 6 | 7 | 3 | 18
  Unknown or Not Reported | 3 | 2 | 4 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Intentions to Lose Weight - Effect of Study Arm on Outcomes
Description: Intention to lose 10lbs in the next 6 months was measured on a 5-point likert scale (1-strongly disagree;5-strongly agree). Responses were examined by study arm.
Time Frame: 3 months after viewing obesity risk assessment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- No Risk Feedback: Control - no obesity risk feedback provided.
- Genetic and Lifestyle Risk Feedback: FTO variant: Relative risk estimates presented based on individuals' risk for obesity from genotype results.
  Lifestyle: Relative risk estimates presented based on individuals' risk for obesity due to personal lifestyle factors (specifically, hours sitting while watching TV).
Arm/Group | No Risk Feedback | Genetic Risk Feedback | Lifestyle Risk Feedback | Genetic and Lifestyle Risk Feedback
Number analyzed (Participants) | 167 | 180 | 177 | 172
units on a scale | 3.06 [2.93 to 3.19] | 3.37 [2.24 to 3.50] | 3.26 [3.13 to 3.39] | 3.26 [3.13 to 3.39]
Statistical Analysis 1: Comparison: No Risk Feedback vs Genetic Risk Feedback vs Lifestyle Risk Feedback vs Genetic and Lifestyle Risk Feedback; Test type: Superiority or Other; p = .0150, Regression, Linear; Adjusted for age, gender, BMI, baseline intention

2. Primary Outcome: Intention to Lose Weight - Impact of Risk Status
Description: Intention to lose 10lbs in the next 6 months measured on a 5-point likert scale (1-strongly disagree;5-strongly agree). This was examined by study arm and level of feedback received (high or elevated risk vs low or non-elevated risk).
Time Frame: 3 months after viewing obesity risk assessment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Low Genetic Risk Feedback: Genetic feedback arm; did not have elevated risk for obesity based on FTO alone.
- High Genetic Risk Feedback: Genetic feedback arm; had elevated risk for obesity based on FTO alone.
- Low Lifestyle Risk Feedback: Lifestyle feedback arm; did not have elevated risk for obesity based on lifestyle behavior alone.
- High Lifestyle Risk Feedback: Lifestyle feedback arm; had elevated risk for obesity based on lifestyle behavior alone.
Arm/Group | No Risk Feedback | Low Genetic Risk Feedback | High Genetic Risk Feedback | Low Lifestyle Risk Feedback | High Lifestyle Risk Feedback
Number analyzed (Participants) | 167 | 69 | 111 | 54 | 123
units on a scale | 3.05 [2.91 to 3.19] | 3.38 [3.17 to 3.59] | 3.35 [3.18 to 3.52] | 3.38 [3.15 to 3.61] | 3.19 [3.03 to 3.36]
Statistical Analysis 1: Comparison: No Risk Feedback vs Low Genetic Risk Feedback vs High Genetic Risk Feedback vs Low Lifestyle Risk Feedback vs High Lifestyle Risk Feedback; Test type: Superiority or Other; p = 0.0365, Regression, Linear; Adjusted for age, gender, BMI, and baseline intent

3. Primary Outcome: Intention to Lose Weight - Combined Risk
Description: Intention to lose 10lbs in the next 6 months on a 5-point likert scale (1-strongly disagree; 5-strongly agree). This was examined by study arm and by combined levels of feedback (e.g. elevated genetic risk and non-elevated lifestyle risk)
Time Frame: 3 months from viewing obesity risk assessment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Low Genetic Risk + Low Lifestyle Risk Feedback: Feedback received: Did not have elevated risk for obesity based on FTO; did not have elevated risk for obesity based on lifestyle behavior.
- Low Genetic Risk + High Lifestyle Risk Feedback: Feedback received: Did not have elevated risk for obesity based on FTO; had elevated risk for obesity based on lifestyle behavior.
- High Genetic Risk + Low Lifestyle Risk Feedback: Feedback received: Had elevated risk for obesity based on FTO; did not have elevated risk for obesity based on lifestyle behavior.
- High Genetic Risk + High Lifestyle Risk Feedback: Feedback received: Had elevated risk for obesity based on FTO; Had elevated risk for obesity based on lifestyle behavior.
Arm/Group | No Risk Feedback | Low Genetic Risk + Low Lifestyle Risk Feedback | Low Genetic Risk + High Lifestyle Risk Feedback | High Genetic Risk + Low Lifestyle Risk Feedback | High Genetic Risk + High Lifestyle Risk Feedback
Number analyzed (Participants) | 167 | 20 | 43 | 33 | 76
units on a scale | 3.08 [2.96 to 3.21] | 3.38 [3.03 to 3.72] | 3.12 [2.88 to 3.36] | 3.24 [2.97 to 3.51] | 3.37 [3.19 to 3.56]
Statistical Analysis 1: Comparison: No Risk Feedback vs Low Genetic Risk + Low Lifestyle Risk Feedback vs Low Genetic Risk + High Lifestyle Risk Feedback vs High Genetic Risk + Low Lifestyle Risk Feedback vs High Genetic Risk + High Lifestyle Risk Feedback; Test type: Superiority or Other; p = 0.0622, Regression, Linear; Adjusted for age, gender, BMI, and baseline intent

ADVERSE EVENTS:
Time Frame: 1 year, 11 months
Groups:
- No Risk Feedback: Control arm - no obesity risk feedback provided
- Genetic Risk Feedback: FTO variant: Relative risk estimates will be presented based on individuals'risk for obesity based on genotype results.
- Both Genetic and Lifestyle Risk Feedback: FTO variant: Relative risk estimates will be presented based on individuals'risk for obesity based on genotype results.
  Lifestyle: Relative risk estimates will be presented based on individuals' risk for obesity due to lifestyle factors.
Arm/Group | No Risk Feedback | Genetic Risk Feedback | Lifestyle Risk Feedback | Both Genetic and Lifestyle Risk Feedback
Serious Adverse Events (participants affected / at risk) | 0/198 | 0/203 | 0/196 | 0/201
Other Adverse Events (participants affected / at risk) | 0/198 | 0/203 | 0/196 | 0/201

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No